CLINICAL TRIAL: NCT02040883
Title: Phase 4 Study of Efficacy and Safety of Tandospirone Combined With Atypical Antipsychotic Drugs to Improve Cognitive Function in Schizophrenia
Brief Title: Tandospirone Combined With Atypical Antipsychotic Drugs in Schizophrenia
Acronym: TAAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qingyun Yin (Other Government)
Responsible Party: Sponsor-Investigator, Qingyun Yin, Professor, Guangzhou Psychiatric Hospital
Organization: Guangzhou Psychiatric Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSPC-SED20130516
Record Dates: First submitted 2014-01-14; First posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Tandospirone; Cognitive Therapy
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; tandospirone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Treated with a stable dose of an AAPD for at least three months before enrollment; Atypical antipsychotic drugs(AAPDs): Risperidone/Olanzapine/Quetiapine/Ziprasidone/Aripiprazole
  Interventions: Drug: Risperidone/Olanzapine/Quetiapine/Ziprasidone/Aripiprazole
- Study Group (Experimental): Atypical antipsychotic drugs(AAPDs) and Tandospirone ; Atypical antipsychotic drugs(AAPDs) ,treated with a stable dose of an AAPD for at least three months before enrollment; AAPD: Risperidone/Olanzapine/Quetiapine/Ziprasidone/Aripiprazole; Tandospirone, 30mg per day;
  Interventions: Drug: Risperidone/Olanzapine/Quetiapine/Ziprasidone/Aripiprazole; Drug: Tandospirone

INTERVENTIONS:
Drug: Risperidone/Olanzapine/Quetiapine/Ziprasidone/Aripiprazole — Treated with a stable dose of an AAPD for at least three months before enrollment, which is suggested to attain the stable cognitive status.
  Other Names: AAPD
Drug: Tandospirone — Tandospirone，30mg per day
  Other Names: Sediel
  Arms: Study Group

SUMMARY:
Efficacy and safety of Tandospirone combined with Atypical Antipsychotic drugs to Improve Cognitive function in Schizophrenia

DETAILED DESCRIPTION:
With atypical antipsychotics for the control group, evaluate cognitive function in schizophrenia patients with antipsychotics combined 5-Hydroxytryptamine 1A (5-HT1A) receptor partial agonist tandospirone

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders-IV Edition (DSM-IV) diagnostic criteria for schizophrenia patients.
* 18-65 years (including 18 and 65), male or female.
* Treated with a stable dose of an AAPD for at least three months.
* Informed consent was obtained (if the patient is in the acute phase of schizophrenia, does not have the capacity, their guardians need sign informed consent).
* PANSS negative score ≤60.

Exclusion Criteria:

* Combined AxisⅠmental illness other than schizophrenia;
* Taking a mood stabilizer, antidepressants, anticholinergic or anxiolytic drugs, and other drugs improve cognitive function;
* Suicidal tendencies;
* Have severe or unstable heart, liver, kidney, endocrine, blood and other medical disease patients
* Clinically significant ECG or laboratory abnormalities were
* Glaucoma and epilepsy;
* Unsupervised or unable to take prescribed medication;
* History of alcohol and drug abuse;
* Allergic;
* Pregnant or lactating woman;
* Patients participate in other clinical trials during a month;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Measurement and treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery(MCCB) total score | From baseline to 12 weeks of treatment

SECONDARY OUTCOMES:
MATRICS Consensus Cognitive Battery(MCCB) factor score | From baseline to 12 weeks of treatment
Positive and Negative Syndrome Scale(PANSS) total score | From baseline to 12 weeks of treatment
Positive and Negative Syndrome Scale(PANSS) factor score | From baseline to 12 weeks of treatment
Personal and Social Performance Scale(PSP) total score | From baseline to 12 weeks of treatment
Clinical Global Impression(CGI) factor score | From baseline to 12 weeks of treatment
Treatment Emergent Symptom Scale(TESS) factor score | From baseline to 12 weeks of treatment
Functional magnetic resonance imaging(FMRI) | From baseline to 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Qingyun Yin, Principal Investigator — Guangzhou Psychiatric Hospital
Locations (1):
- Guangzhou Psychiatric Hospital, Guangzhou, Guangdong, China